CLINICAL TRIAL: NCT03783585
Title: Assessment of the Feasibility of a Web-based CBT-I Intervention to Improve Sleep Quality and Fatigue in Individuals With Multiple Sclerosis
Brief Title: Feasibility of Web-based CBT-I Intervention in Individuals With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Catherine Siengsukon, PT, PhD, Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00142464
Record Dates: First submitted 2018-10-01; First posted 2018-12-21 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive behavioral therapy for insomnia (CBT-I) (Experimental): Participants randomized to this arm will participate in a 6-week web-based cognitive behavioral therapy for insomnia (CBT-I) program.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia
- CBT-I + biweekly support (Experimental): Participants randomized to this arm will participate in a 6-week web-based CBT-I program. In addition, biweekly support consisting of one-on-one, semi-structured, online video-chat sessions (via HIPAA-compliant Zoom) or phone calls will be conducted every other week.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia; Behavioral: Cognitive behavioral therapy for insomnia + biweekly support

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia — The web-based CBT-I program is a 6-week interactive, online program that delivers typical CBT-I treatment techniques of stimulus control, sleep restriction, behavioral modifications, and cognitive restructuring.
Behavioral: Cognitive behavioral therapy for insomnia + biweekly support — Individuals randomized into the CBT-I + biweekly support will participate in CBT-I as described as well as a biweekly phone call or video call with research personnel for motivational interviewing.
  Arms: CBT-I + biweekly support

SUMMARY:
Forty individuals with multiple sclerosis (MS) will be randomly assigned to a 6-week web-based cognitive behavior therapy for insomnia intervention (wCBT-I) or to wCBT-I plus biweekly support meetings with research personnel via phone or video. Questionnaires will be used to assess sleep quality, fatigue, and satisfaction. Recruitment, retention, attrition, adherence, and safety information will also be collected. This study is significant because addressing insomnia symptoms through CBT-I could be a low-cost, low-risk, non-pharmacological options for improving sleep quality and MS symptoms in individuals with MS. This study is innovative because CBT-I has never been delivered via a web-based application to individuals with MS which may increase access to services.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* diagnosis of MS by physician
* report of difficulty falling asleep, maintaining sleep, or waking up too early at least 3 nights/week for the past 6 months
* ≥10 on Insomnia Severity Index (ISI)
* English speaking
* reports access to internet service and phone
* has a high school diploma to serve as a proxy measurement of reading ability to ensure adequate reading ability to participate in the study.

Exclusion Criteria:

* known untreated sleep disorder (such as sleep apnea or restless leg syndrome)
* >3 on STOP BANG indicating risk of sleep apnea
* increased risk of restless leg syndrome
* nervous system disorder other than MS
* relapse and/or corticosteroid use in past 8 weeks
* score of ≥15 on the Patient Health Questionnaire (PHQ-9) indicating severe depression or endorse any suicidal ideation (answer 1, 2 or 3 on #9 of the PHQ-9)
* performs shift-work.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
change in Insomnia Severity Index (ISI) | baseline and week 8
  The ISI is a valid and reliable measure of sleep difficulties and consists of 7 questions each rated on a 0-4 scale. The range of scores on the ISI is 0-28, with ≥10 suggesting clinical insomnia

SECONDARY OUTCOMES:
change in Pittsburgh Sleep Quality Index (PSQI) | baseline and week 8
  The PSQI is a well-validated and reliable measure of sleep quality and consists of 9 items within 7 sleep categories. The 7 sleep category scores are summed to form a single global score ranging from 0-21. A global score of >5 reflects poor sleep quality
change in Modified Fatigue Impact Scale (MFIS) | baseline and week 8
  The MFIS consists of 21 items with 3 subscales: physical, cognitive, and psychosocial. The score on the 21 items are scored with a range of 0-84 with a higher score indicating a greater impact of fatigue.
change in Fatigue Severity Scale (FSS) | baseline and week 8
  Fatigue Severity Scale (FSS) assesses the impact of fatigue on activities for the week prior and consists of 9 questions. The mean of the 9 scores is calculated with a range of 0-7.
change in Multiple Sclerosis Impact Scale (MSIS) | baseline and week 8
  MSIS-29 is total of 29 items scale, with subscales of physical (20 items) and psychological (9 items). Responses computed in a range from 0-100, and higher scores indicating a worse quality of life due to physical and physiological impacts of MS.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Siengsukon, PT, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Catherine Siengsukon, Kansas City, Kansas, United States